CLINICAL TRIAL: NCT04157361
Title: Pulmonary Condensate: A Promising Source of Proteomic Biomarkers for Non-invasive Evaluation of Pulmonary Involvement in Asthma and Cystic Fibrosis.
Brief Title: Pulmonary Condensate: Non-invasive Evaluation of Pulmonary Involvement in Asthma and Cystic Fibrosis.
Status: Recruiting | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Sponsor
Other Study IDs: 122
Record Dates: First submitted 2019-10-11; First posted 2019-11-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Bronchial Asthma; Pulmonary Cystic Fibrosis
Keywords: Breath condensate; Bronchial asthma; Cystic Fibrosis
MeSH Terms: conditions — Asthma; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath condensate, serum and blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asthma: Children/adults with moderate or IgE mediated asthma with inhaled and/or food allergies before and during inhaled corticosteroid, leukotriene modifiers or long-acting beta agonists treatment.
  Interventions: Diagnostic Test: Collection of breath condensate
- Cystic fibrosis: Children/adults with cystic fibrosis before and after antibiotics treatment and during clinical deterioration.
  Interventions: Diagnostic Test: Collection of breath condensate
- Healthy control: Healthy control children/adults without chronic or autoimmune disease
  Interventions: Diagnostic Test: Collection of breath condensate

INTERVENTIONS:
Diagnostic Test: Collection of breath condensate — Breath condensate will be collected from the patients involved in study.

SUMMARY:
Exhaled breath condensate (EBC) represents a rich source for countless biomarkers that can provide valuable information about respiratory as well as systemic diseases. Finding non-invasive methods for early detection of lung injury, inflammation and infectious complications in chronic diseases like (CF) Cystic fibrosis or (AB) Bronchial asthma would be highly beneficial. Investigators propose to establish EBC "breathprints" revealing molecular signatures of pulmonary inflammation and specific respiratory bacterial infections of CF patients and AB. Investigators hypothesize that the analysis of EBC can reveal biomarkers specific for severity of the inflammation, and infection caused by opportunistic pathogens such as P. aeruginosa (PA). With these breath-prints, investigators also propose to establish correlations between respiratory microbiota using traditional methods and CF lung disease severity. Together, the studies will advance the development and validation of EBC as a novel tool for the proper diagnosis of AB and monitoring of CF disease activity, treatment efficacy and PA or another opportunistic infections.

DETAILED DESCRIPTION:
Exhaled breath condensate (EBC) represents a rich source for countless biomarkers that can provide valuable information about respiratory as well as systemic diseases. Finding non-invasive methods for early detection of lung injury, inflammation and infectious complications in chronic diseases like Cystic fibrosis (CF) or Bronchial asthma (AB) would be highly beneficial. Investigators propose to establish EBC "breathprints" revealing molecular signatures of pulmonary inflammation and specific respiratory bacterial infections of CF patients and AB. Investigators hypothesize that the analysis of EBC can reveal biomarkers specific for severity of the inflammation, and infection caused by opportunistic pathogens such as P. aeruginosa (PA). With these breath-prints, investigators also propose to establish correlations between respiratory microbiota using traditional methods and CF lung disease severity. Together, the studies will advance the development and validation of EBC as a novel tool for the proper diagnosis of AB and monitoring of CF disease activity, treatment efficacy and PA or another opportunistic infections.

ELIGIBILITY:
Inclusion Criteria:

* Children/adults with moderate or IgE mediated asthma
* Children/adults with cystic fibrosis
* Healthy control children/adults without lung disorders

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with Diagnosis of Cystic Fibrosis
  * Patients with Diagnosis of Asthma
  * Healthy Controls
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker identification using method of High Resolution Mass Spectrometry processed on Orbitrap Velos Elite machine | 18 months from the screening
  Biomarker iidentification in EBC using method of High Resolution Mass Spectrometry in patients with bronchial astma, cystic fibrosis and healthy control.
FEV1 determination in Cystic Fibrosis patients | 18 months from the screening
  Spirometry - FEV1 in Cystic Fibrosis patients and its correlation with biomarker results.
FVC determination in Cystic Fibrosis patients | 18 months from the screening
  Spirometry - FVC in Cystic Fibrosis patients and its correlation with biomarker results.
Amylase readings in blood serum in Cystic Fibrosis patients | 18 months from the screening
  Amylase readings in blood serum in Cystic Fibrosis patients and its correlation with biomarker results.
Lipase readings in blood serum in Cystic Fibrosis patients | 18 months from the screening
  Lipase readings in blood serum in Cystic Fibrosis patients and its correlation with biomarker results.
Microbiology cultivation in Cystic Fibrosis patients | 18 months from the screening
  Sampling for microbiology cultivation and determination of microbes present in EBC, correlation with biomarker results.
CT in Cystic Fibrosis patients | 18 months from the screening
  CT imaging of Cystic Fibrosis patients, correlation with biomarker results.
RTG in Cystic Fibrosis patients | 18 months from the screening
  RTG imaging of Cystic Fibrosis patients, correlation with biomarker results.

SECONDARY OUTCOMES:
Inflamatory biomarker identification using method of High Resolution Mass Spectrometry processed on Orbitrap Velos Elite machine | 18 months from the screening
  Inflamatory biomarker identification in EBC using method of High Resolution Mass Spectrometry in patients with bronchial astma, cystic fibrosis and healthy control.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Dzubak, MD, PhD., Study Director — The Institute of Molecular and Translational Medicine, Czech Republic
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided